CLINICAL TRIAL: NCT00626860
Title: The Use of Dendritic Cell/Tumor Hybridomas as a Novel Tumor Vaccine in Patients With Advance Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, David Avigan, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2001P001112; DCMEL-003-00
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Melanoma
Keywords: melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: DC/tumor fusion vaccine — SC vaccinations administered to each patient at 3-week intervals for 2-3 doses

SUMMARY:
This study aims to determine if the vacccine can be used safely in patients with advanced melanoma (cancer of the pigment cells) and whether the cells in this vaccine are capabale of producing immune responses against your own cancer.

DETAILED DESCRIPTION:
To assess the toxicity associated with vaccination of melanoma patients with dendritic cell (DC)/tumor fusions. To determine if cellular and humoral immunity can be induced by serial vaccination with DC/tumor fusions cells. To determine if vaccination DC/tumor fusions results in a tumor response.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed diagnoses of disseminated melanoma, with measurable and clearly progressive metastatic involevment
* Patients must be at least 18 years old
* Patients must have ECOG performance status 0-1 with greater than 9 week life expectancy
* Those patients with the following accessible tumor will be eligible: soft tissue, bone marrow or visceral lesions; Skin or superficial soft tissue, or lymph nodes amenable to resection under local anesthesia; Patients who require surgical procedures that are not considered significantly invasive but may require general anesthesia, such as thorascopic biopsy, laparascopic biopsy or mediastinal node biopsy may potentially be eligible; Malignant ascites or pleural effusion; Patients requiring major surgical intervention will be considered ineligible. Patients scheduled to undergo tumor resection for independent diagnostic or therapeutic indications may have tumor collected for the purposes of this study.
* Labs: WBC >_ 2.0 x 10x3/uL, Bilirubin <_2.0 mg/dL, Creatine <_ 2.0mg/dL
* Women of childbearing age must have a negative pregnancy test and adequate contraception method(s) must be documented
* All patients must be informed of the investigational nature of this study and must give written informed consent in accordance with institutional and federal guidelines

Exclusion Criteria:

* Patients must not have received other immunotherapy treatment in the past four weeks prior to study entry
* Patients must not have received chemotherapy for three weeks prior to the first vaccination
* Patients must be without evidence of active CNS disease
* Patients must not have clinically significant autoimmune disease
* Patients must be HIV negative
* Patients must not have serious intercurrent illness such as infection requiring IV antibiotics, or significant cardiac disease characterized by significant arrhythmia, ischemic coronary disease or congestive heart failure
* Patients requiring corticosteroids for either melanoma related or co-morbid illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2000-07; Primary Completion 2002-01 (Actual); Study Completion 2008-09-10 (Actual)

PRIMARY OUTCOMES:
To assess the toxicity, cellular and humoral immunity and tumor response in patient with melanoma receiving the DC/tumor fusion vaccine | screening/baseline, treatment period and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: David Avigan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- BIDMC, Boston, Massachusetts, United States